CLINICAL TRIAL: NCT04520802
Title: Neuroinflammation in Cognitive Decline Post-cardiac Surgery: The FOCUS Study
Brief Title: Neuroinflammation in Cognitive Decline Post-cardiac Surgery
Acronym: FOCUS
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Wilson F. Abdo, Principal Investigator, Radboud University Medical Center
Other Study IDs: NL.57785.091.16; 2016-002016-40 (EudraCT Number); CMO 2016-2598 (Other: CMO Regio Arnhem-Nijmegen)
Record Dates: First submitted 2020-07-03; First posted 2020-08-20 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Cognitive Dysfunction; Coronary Artery Disease; Pathophysiology
MeSH Terms: conditions — Postoperative Cognitive Complications; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POCD: Patients with postoperative cognitive decline (POCD) after coronary artery bypass grafting (CABG) surgery
  Interventions: Diagnostic Test: 18F-DPA-714 PET/CT neuroimaging
- no POCD: Patients without postoperative cognitive decline (POCD) after coronary artery bypass grafting (CABG) surgery
  Interventions: Diagnostic Test: 18F-DPA-714 PET/CT neuroimaging

INTERVENTIONS:
Diagnostic Test: 18F-DPA-714 PET/CT neuroimaging — * Pre- and postoperative neuroimaging using 18F-DPA-714 PET/CT and brain MRI.
  * Longitudinal neuropsychological examinations (up to 6 months postoperatively)
  * Blood samples are drawn to assess the severity of the systemic inflammatory response

SUMMARY:
Major cardiovascular surgery is associated with postoperative cognitive decline (POCD), with a deterioration in memory, attention and speed of information processing. A multifactorial pathophysiology is presumed but this study focuses on the role of (neuro)inflammation in the development of POCD after coronary artery bypass grafting (CABG) surgery.

DETAILED DESCRIPTION:
Systemic inflammation can activate the innate immune cells of the brain inducing neuroinflammation, which plays an important role in the pathogenesis of neurodegenerative disease. Major cardiovascular surgery induces a severe systemic inflammatory response.There is growing support that neuroinflammation is a pivotal factor in the development of postoperative cognitive decline (POCD) due to surgery-related systemic inflammation.

Although the neuroinflammatory hypothesis is scientifically accepted, in vivo human data supporting the role of neuroinflammation in severe systemic inflammation such as major surgery are still lacking. In the last decades, several nuclear imaging tracers have been developed that can quantitatively measure microglial and astrocytic activation in vivo, by targeting the mitochondrial 18kDa translocator protein (TSPO).

The investigators hypothesize that cardiac surgery induces a neuroinflammatory response and that its presence is related to acute and long term brain dysfunction postoperatively. This will be studied by pre- and postoperative PET brain imaging using a 18F-DPA-714 tracer targeting TSPO, combined with longitudinal neuropsychological examinations. Structural changes in the brain will be recorded on MRI prior to and after cardiac surgery to enable us to correct for the potentially confounding effects of neurovascular events on cognitive outcomes after CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Planned for on-pump coronary artery bypass grafting surgery
* High-affinity binder or mixed-affinity binders based on rs6971 polymorphism for TSPO
* Chronic use of statins (defined as pre-hospital use)

Exclusion Criteria:

* Previous cardiac surgery.
* Pregnancy or wish to become pregnant within 2 weeks after PET-CT scan
* Contra-indication to undergo a PET/CT or MRI scan, including claustrophobia.
* Low-affinity binder based on rs6971 polymorphism for TSPO, or unable to determine rs6971 polymorphism.
* Patients with cognitive disorders that have not recovered enough to be able to understand the study leaflets and information for participation.
* Brain or spinal surgery within the last 6 months.
* Meningitis or brain infection within the last 6 months.
* Pre-existing dementia or neurodegenerative disease or cognitive impairment interfering with the ability to understand informational material about this research project.
* Presence of a CSF catheter or shunt.
* Patients with known brain tumors.
* Patients with brain injury (e.g. acute stroke, or subarachnoid hemorrhage) within the last 6 months.
* Severe brain trauma in previous medical history.
* Chronic (>2 weeks) use of immunosuppressive agents (see table 3.3.A).
* Concomitant diseases resulting in severe immunosuppression (e.g. HIV).
* Auto-immune or auto-inflammatory disease
* Active infection < 2 weeks prior to inclusion (defined as fever >38.5 or antibiotic treatment)
* Kidney failure, defined by a MDRD-GFR<15 ml/min/1.73m2
* Known contrast allergy for gadolinium
* Chronic use of neuroleptics, defined as pre-hospital use.
* Patients that do not speak Dutch or have disabilities that prevent accurate delirium diagnosis.
* Analphabetic patients.
* No written informed consent obtained.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients >50 years that are planned to undergo elective coronary artery bypass grafting (CABG) surgery by the cardiothoracic surgery department of the Radboud university medical center in Nijmegen (NL).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in TSPO PET tracer uptake at 3-7 days post-surgery | 3-7 days post-surgery minus preoperative (= day before surgery)
  18F-DPA-714

SECONDARY OUTCOMES:
Occurrence of postoperative cognitive dysfunction (POCD) | Baseline (preoperative), postoperative (3-7 days after surgery, 6 weeks and 6 months)
  POCD diagnosis based on neuropsychological assessments including TMT A&B, Stroop I, II, III, WAIS-IV - digit span, LDST, RAVLT, RCFT, RBMT-3 face recognition, LFT and token test. POCD diagnosis is made when patients are newly impaired in one or more cognitive domains (memory, executive functioning, speed of processing and language), or when the average test rating has declined in more than one domain compared to baseline.
Whole brain TSPO PET tracer uptake pre- and 3-7 days post-surgery | pre- and 3-7 days post-surgery
  18F-DPA-714
Pro- and anti-inflammatory in vivo cytokine concentrations [in pg/ml] | Day before surgery, during surgery (stop extracorporeal circulation (ECC)), after surgery (6 hours after stop ECC, 24 hours after incision, 3-7 days post-surgery and 6 weeks after surgery)
  TNFa, IL6, IL-1B, IL10, IL-1RA
Ex vivo cytokine production of stimulated monocytes [in ng/10^9 monocytes] | Day before surgery, 3-7 days and 6 weeks after surgery
  TNFa, IL6, IL1B, MCP1, IL10
Flowcytometry analysis to study the inflammatory phenotype of the cells | Day before surgery, 3-7 days and 6 weeks after surgery
  HLA-DR, CCR2, CD11b, CD14, CD16
Complete blood count | Day before surgery, during surgery (stop extracorporeal circulation (ECC)), after surgery (6 hours after stop ECC, 24 hours after incision, 3-7 days post-surgery and 6 weeks after surgery)
  including leukocyte differentiation measured on an automated hematology analyzer
Ex vivo cytokine production of healthy donor monocytes, after exposure to patient serum obtained during CABG surgery | Perioperatively at stop extracorporeal circulation (ECC)
  Healthy donor monocytes will be exposed to patient serum obtained during surgery, to see whether this changes the ex vivo cytokine producing capacity (TNFa, IL6, IL10)
Number of newly developed (ischemic and hemorrhagic) brain and vascular wall lesions | pre- and 3-7 days post-surgery
Delta brain activity in three large scale brain networks involved in stress reactivity on resting-state fMRI | pre- and 3-7 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wilson F Abdo, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Department of Intensive Care Medicine, Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peters van Ton AM, Duindam HB, van Tuijl J, Li WW, Dieker HJ, Riksen NP, Meijer FA, Kessels RP, Kohn N, van der Hoeven JG, Pickkers P, Rijpkema M, Abdo WF. Neuroinflammation in cognitive decline post-cardiac surgery (the FOCUS study): an observational study protocol. BMJ Open. 2021 May 11;11(5):e044062. doi: 10.1136/bmjopen-2020-044062. PMID 33980522
- See also: Pubmed link to publication of complete study protocol — https://pubmed.ncbi.nlm.nih.gov/33980522/